CLINICAL TRIAL: NCT02367911
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis
Brief Title: A Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122-0551-305
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Experimental): 122-0551 Foam, topically applied twice daily for two weeks
  Interventions: Drug: 122-0551 Foam
- Vehicle Arm (Placebo Comparator): Vehicle Foam, topically applied twice daily for two weeks
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: 122-0551 Foam — 122-0551 Foam applied twice daily to treat psoriasis
  Arms: Active Arm
Drug: Vehicle Foam — Vehicle Foam applied twice daily to treat psoriasis
  Arms: Vehicle Arm

SUMMARY:
This Phase 3 study has been designed to determine and compare the efficacy and safety of 122-0551 Foam and Vehicle Foam applied twice daily for two weeks in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than 12% affected body surface area.
* Subject has an Investigator's Global Assessment (IGA) score of at least three (moderate) at study start.
* If subject is a woman of childbearing potential, she must have a negative urine pregnancy test and agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
* Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, or which exposes the subject to an unacceptable risk by study participation.
* Subject has used any phototherapy (including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days prior to study start.
* Subject has used any systemic methotrexate, retinoids, systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids], cyclosporine or analogous products within 90 days prior to study start.
* Subject has used any systemic biologic therapy (i.e., FDA-approved or experimental therapy) within five half-lives of the biologic prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Andrasfay, Study Director — Therapeutics, Inc.
Locations (9):
- United States (9):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - UCSD Dermatology, San Diego, California
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Dermatology Consulting Services, High Point, North Carolina
  - Arlington Research Center, Inc., Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2015 to August 2015
  The location of clinical sites included dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Period: Overall Study
Arm/Group | Active Arm | Vehicle Arm
Started | 71 | 73
Completed | 66 | 69
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline demographics is based on the Intent-To-Treat (ITT) population, defined as all enrolled subjects in the study who were randomized and dispensed the test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Vehicle Arm | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.44) | 52.0 (13.75) | 52.2 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 66 | 69 | 135
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 2 | 3
  Race: Black or African American | 2 | 7 | 9
  Race: White | 68 | 64 | 132
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 73 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Rated a "Treatment Success" Based on the Investigator's Global Assessment (IGA)
Description: The IGA score is a static evaluation of the overall or "average" degree of severity of a subject's disease, taking into account all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. IGA is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Time Frame: Day 15
Population: Analysis shown is based on the ITT population, defined as all enrolled participants who were randomized and dispensed the test article.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 71 | 73
percentage of participants | 18.3 | 9.6

2. Secondary Outcome: Percentage of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: A static assessment of the overall or "average" degree of severity of each of three key characteristics present within all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. Each clinical sign of psoriasis is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 15
Population: Analysis shown is based on the Intent-to-Treat (ITT) population, defined as all enrolled participants who were randomized and applied at least one dose of the test article. Missing data was imputed as failure.
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm | Vehicle Arm
Number analyzed (Participants) | 71 | 73
percentage of participants
  Scaling | 32.4 | 13.7
  Erythema | 16.9 | 8.2
  Plaque Elevation | 26.8 | 13.7

3. Other Pre Specified Outcome: Proportion of Subjects With IGA "Treatment Success"
Description: "Treatment success" and IGA as defined in the primary outcome measure.
Time Frame: Day 8
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Proportion of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: "Treatment success" and clinical signs as defined in the secondary outcome measure.
Time Frame: Day 8
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change From Baseline in Pruritus Score
Description: Pruritus scale will be used to assess the subjective and multidimensional experience of the subject's pruritus (itching) during the previous two weeks at Baseline and Day 15. Possible scores range from 5 (no pruritus) to 25 (most severe pruritus).
Time Frame: Day 15
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in % Body Surface Area (BSA) With Active Psoriasis
Description: The investigator will use the assumption that 1% BSA is approximately equal to the surface area of the subject's palm and fingers, with the fingers extended yet grouped together, creating a flat oval-like surface area.
Time Frame: Day 8 and Day 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events (AEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 15) or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The safety population included all participants enrolled in the study who were dispensed and applied the test article at least once; because the first dose of the test article was applied at the study site (Day 1), all participants (N=144) were included in the safety population.
Arm/Group | Active Arm | Vehicle Arm
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 2/71 | 3/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=71) | Vehicle Arm (N=73)
Application site dryness (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review thirty days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.